CLINICAL TRIAL: NCT05492370
Title: Effects of a Yeast Fermentate (EpiCor) Supplement on Cold or Flu Symptoms in Healthy Children: A Randomized, Double-blind, Placebo Controlled Clinical Trial
Brief Title: Effects of a Yeast Fermentate (EpiCor) Supplement on Cold or Flu Symptoms in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21CLRFZ02
Record Dates: First submitted 2022-07-29; First posted 2022-08-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Signs and Symptoms, Respiratory
MeSH Terms: conditions — Signs and Symptoms, Respiratory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EpiCor (Experimental): 500 mg EpiCor given as two gummy supplements. Participants will be instructed to take two gummies per day in the morning, with or without food, for 84 days, starting on Day 1.
  Interventions: Dietary Supplement: EpiCor
- Placebo (Placebo Comparator): Two gummy supplements. Participants will be instructed to take two gummies per day in the morning, with or without food, for 84 days, starting on Day 1.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EpiCor — 2 gummies daily
  Arms: EpiCor
Dietary Supplement: Placebo — 2 gummies daily
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled study. The purpose of the clinical study is to determine the difference between 84 days of once daily oral EpiCor supplementation compared to placebo on the incidence of cold or flu symptoms among children aged 4-12 years who are attending school or daycare.

DETAILED DESCRIPTION:
This double-blind, randomized, placebo-controlled study aims to determine the difference between 84 days of once daily oral EpiCor supplementation compared to placebo on the incidence of cold or flu symptoms among children aged 4-12 years who are attending school or daycare. Healthy children, with parental consent, are included in the study. The study includes one screening visit (day -45 to -15), a run-in period (day -14 to -1), and 3 clinical visits: day 0 (baseline), day 42, and day 84 (end of study). During the screening visit, the investigator reviews medical history, concomitant therapies, current health status, assesses inclusion and exclusion criteria, vital signs, weight and height measurements, assesses pre-emergent adverse events, and dispenses saliva collection kit for salivary Immunoglobulin A (IgA) analysis as well as study dairy and Canadian Acute Respiratory Illness and Flu Scale (CARIFS) questionnaire. Participants complete the CARIFS questionnaire and study dairy during the run-in period. On day 0, participants return to the clinic with their saliva collecting kit, completed study diaries, and CARIFS questionnaire for baseline assessments; during this visit, eligible participants are randomized and they are also instructed to initiate investigational product administration on the morning of day 1. At day 42, participants and their caregivers return to the clinic for assessments with unused investigation product, saliva collection kit, completed study diaries, CARIFS questionnaire, and a Questionnaire for measuring health-related Quality of Life in Children and Adolescents (KINDL); investigator reviews concomitant therapies and adverse events, dispenses new study diary, CARIFS questionnaire, saliva collection kit, investigational product, and measures vital signs, weight, and height. The same procedure is repeated during the last clinical visit at day 84 (end of study), except that no investigational product is provided. Daily throughout the study, participant caregivers complete the study diary to track missed school or daycare days, well days, use of prescription/non-prescription cold/flu medication, adverse events, and concomitant therapies, and cold or flu symptoms (via CARIFS questionnaire when cold or flu symptoms are present).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the age of 4-12 years of age, inclusive
* Individuals of child-bearing potential must have a negative baseline urine pregnancy test
* Enrolled in and attending school or daycare at baseline
* Healthy as determined by medical history and review of health status as per Qualified Investigator
* Agrees to maintain current lifestyle habits as much as possible throughout the study depending on their ability to maintain the following: diet, medications, supplements, exercise, and sleep and avoid taking new supplements
* Willing to complete evaluations, measurements, questionnaires, diaries, and tests associated with each clinic visit and be compliant to study product intake throughout the study
* A care provider who can reliably bring the participant to all study visits; the participant's primary caregiver must be willing and able to complete the questionnaires
* The child and the child's parent(s) or legal guardian(s) have given voluntary, written, informed consent to partake in the study

Exclusion Criteria:

* Individuals who are pregnant
* Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients
* History or presence of a clinically relevant cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal condition which affects absorption, or pancreatic disorders, as assessed by the Qualified Investigator
* Immune dysfunction and/or taking an immunosuppressive medication
* Severe environmental allergies requiring medication or need for allergy shots
* Cancer. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
* Asthma, as assessed by the Qualified Investigator
* Participants with siblings that live in the same household and are eligible for the study unless they are enrolled consecutively (e.g., not enrolled at the same time)
* Participation in a clinical research trial within 30 days prior to randomization, as assessed by the Qualified Investigator
* Participant or participant's caregiver who are cognitively or neurodevelopmentally impaired and/or are unable to give informed consent
* Any other condition that may adversely affect the ability to complete the study or its measures or which may pose significant risk to the participant as assessed by the Qualified Investigator

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Incidence of cold or flu symptoms | 84 days
  To determine the difference between 84 days of once daily oral EpiCor supplementation compared to placebo on the incidence of cold or flu symptoms among children aged 4-12 years who are attending school or daycare.

SECONDARY OUTCOMES:
Incidence on cold or flu symptoms from baseline to day 42 | 42 days
  Determine the difference between EpiCor and placebo from baseline to day 42 on the incidence of cold or flu symptoms during an 84-day supplementation period
Severity of cold or flu symptoms | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84, assessed of the individual items on CARIFS and by area under the curve (AUC) for the CARIFS daily symptom score. The CARIFS questionnaire includes 18 items answered on a 4-point scale (no problem = 0, minor problem = 1, moderate problem = 2, major problem = 3) across three domains (symptoms, function, and parental impact). The higher the score, the more sever the illness.
Duration of cold or flu symptoms | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84
Proportion of children with no cold or flu symptoms | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84
Number of days prior to first cold or flu symptoms | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84
Number of missed school or daycare days due to cold or flu symptoms | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84
Number of well days, related to the absence of cold or flu symptoms | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84
Use of prescription and non-prescription cold/flu medications to treat cold or flu symptoms | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84
Saliva secretory immunoglobulin A concentrations | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84
Quality of life as assessed by the KINDL questionnaire | At 42 and 84 days
  To determine the difference between EpiCor compared to placebo from baseline to day 42 and to day 84. The KINDL questionnaire will be used to assess quality of life. This questionnaire contains 46 questions (scored 1-5; 1 - never, 2 - seldom, 3 - sometimes, 4 - often, 5 - all the time) answered by the caregiver.
Safety profile as assessed by Adverse Events (AEs) | At 42 and 84 days
  To determine EpiCor safety profile in children aged 4-12 years as assessed by AEs for 42 and 84 days.
Safety profile as assessed by vital sign blood pressure | At 42 and 84 days
  To determine EpiCor safety profile in children aged 4-12 years as assessed by blood pressure for 42 and 84 days.
Safety profile as assessed by vital sign heart rate | At 42 and 84 days
  To determine EpiCor safety profile in children aged 4-12 years as assessed by heart rate for 42 and 84 days.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science
Locations (1):
- KGK Science Inc, London, Ontario, Canada